CLINICAL TRIAL: NCT01818583
Title: Potassium Infusion for Conversion of Atrial Fibrillation/-Flutter
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Kiarash Tazmini, Kiarash Tazmini, MD, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AK-01
Record Dates: First submitted 2013-03-22; First posted 2013-03-26 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial fibrillation; Atrial flutter; Potassium; Cardioversion
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Potassium Chloride; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Potassium (Experimental): Potassium chloride infusion at a rate of 15 mmol/h (60 mmol KCl in 1000 ml of 5% glucose with a concentration of 0.05 mmol/mL, flow rate 265 mL/h). If the serum Mg ≤0.8 mmol/L, MgSO4 infusion (0.5 mmol/kg/24 hours in 1000 mL NaCl 0.9% corresponding to an infusion rate of approximately 42 mL/hour) will also be administered.
  Interventions: Drug: Potassium chloride
- Placebo (Placebo Comparator): 5% glucose (flow rate 265 ml/h) as placebo infusion.
  Interventions: Drug: Glucose 50 MG/ML

INTERVENTIONS:
Drug: Potassium chloride
  Arms: Potassium
Drug: Glucose 50 MG/ML
  Arms: Placebo

SUMMARY:
Atrial fibrillation is a condition in which the heart's upper chambers, the atria, contract at an abnormally rapid rate. It is a common type of arrhythmia, and occurs in 1-2% of the general population. The prevalence of atrial fibrillation increases with age. Between 50 and 70% of patients with atrial fibrillation lasting <48 hours spontaneously convert to normal sinus rhythm, and drug therapy increases the likelihood of conversion to sinus rhythm. Another treatment option for conversion of atrial fibrillation and atrial flutter is electrical conversion. This is an effective treatment but requires anesthesia.

Current treatment strategy for medical conversion of atrial fibrillation and atrial flutter is to employ drugs that affect ion channel activity in atrial cardiomyocytes. However, such converting drugs all have potentially serious side effects and are expensive. Potassium, sodium, calcium, and magnesium molecules are the most important ions causing electric current in the heart tissue. Our hypothesis is that hypokalemia promotes atrial fibrillation/atrial flutter by a direct effect on cardiomyocytes. Accordingly, we also hypothesize that potassium infusion may convert atrial fibrillation/atrial flutter to normal sinus rhythm. If so, this would be an inexpensive treatment with potentially very few side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal atrial fibrillation/atrial flutter with duration <48 hours
* Plasma potassium ≤4,0 mmol/L.
* Age ≥ 18 år

Exclusion Criteria:

* Plasma potassium > 4,0 mmol/L
* eGFR <30 mL/min
* Patients on antiarrhythmic therapy (flecainid, amiodarone, dronedarone or sotalol)
* Pregnancy
* Breast feeding
* Patients participating in a clinical trial during the last six months
* Addison disease, adynamia episodic hereditary, or Sickle cell anemia
* Metabolic acidosis, pH < 7,2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Cardioversion (time and percentage) | 24 hours

SECONDARY OUTCOMES:
Atrial fibrillation at 3 months follow up visit and during 72 hours ECG-monitoring period. | At about 3 months follow up, plus additional 3 days ECG-monitoring
  The patients will be followed up with a resting ECG about three months after study intervention, and subsequently on-demand ECG will be monitored for 72 hours.

OTHER OUTCOMES:
Adverse events | During time of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Erik Øie, MD, PhD, Study Director — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tazmini K, Fraz MSA, Nymo SH, Stokke MK, Louch WE, Oie E. Potassium infusion increases the likelihood of conversion of recent-onset atrial fibrillation-A single-blinded, randomized clinical trial. Am Heart J. 2020 Mar;221:114-124. doi: 10.1016/j.ahj.2019.12.014. Epub 2019 Dec 27. PMID 31986288